CLINICAL TRIAL: NCT02819401
Title: A Prospective, Open-label, Post-marketing Observational Study to Evaluate the Effects of High-fiber Enteral Pediatric Formula in Children With Failure to Thrive Due to Malnutrition
Brief Title: The Effects of a High-fiber Formula in Children With Failure to Thrive
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: ANTK1001
Record Dates: First submitted 2016-03-18; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: GI Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: pediatric formula — high-fiber enteral formula

SUMMARY:
The present study is designed to determine the gastrointestinal tolerability of enteral nutritional products, physicians and parents' overall perception of enteral nutrition products as well as providing basic demographic information on pediatric populations prescribed these formula for supportive treatment as part of the routine healthcare service in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Age; 1-10 years (inclusive)
* Children diagnosed as failure-to-thrive(FTT).
* Children who have been recently prescribed and treatment initiated with isocaloric or hypercaloric high-fiber pediatric enteral formula suitable for oral and/or nasogastric tube feeding before inclusion in the study.

Exclusion Criteria:

* Chronic renal disorder
* Decompensated liver disease
* Any other chronic condition that was not under control (e.g. diabetes, thyroid disorder, etc.)
* Any type of malignant disease including leukemia and lymphoma
* Cystic fibrosis
* Short bowel syndrome
* Any type of food allergy or intolerance
* Growth hormone deficiency
* Use of enteral feeding within the last 4 weeks

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with failure to thrive who are receiving a high-fiber enteral formula for supportive treatment as part of the routine healthcare service in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Physician Perception of Formula Use | Baseline to Month 6
  Questionnaire

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Baseline to Month 1, Month 2, Month 4 and Month 6
  Subject questionnaires
Description of Population | Baseline
  Demographic collection of patients recommended high-fiber enteral formula
Weight | Baseline to Month 1, Month 2, Month 4 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Aysugul Alptekin, MD, Study Chair — Abbott Turkey
Locations (17):
- Turkey (Türkiye) (17):
  - Ankara Üniversitesi Tıp Fakültesi, Ankara
  - Trakya Üniversitesi Tıp Fakültesi, Edirne
  - Fırat Üniversitesi Tıp Fakültesi, Elâzığ
  - Özel Doğu Anadolu Hastanesi, Elâzığ
  - Gaziantep Üniversitesi Tıp Fakültesi, Gaziantep
  - Memorial Şişli Hastanesi, Istanbul
  - Medeniyet Üniversitesi Göztepe Eğitim ve Araştırma Hastanesi, Istanbul
  - Dr.Sadi Konuk Eğitim ve Araştırma Hastan, Istanbul
  - Şifa Üniversitesi Bornova Sağlık Uygulama ve Araştırma Merkezi, Izmir
  - Behçet Uz Çocuk Hastalıkları Hastanesi, Izmir
  - İzmir Tepecik Eğitim ve Araştırma Hastanes, Izmir
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri̇
  - Kocaeli Üniversitesi Tıp Fakültesi, Kocaeli
  - Konya Üniversitesi Selçuk Tıp Fakültesi, Konya
  - Kırıkkale Üniversitesi Tıp Fakültesi, Kırıkkale
  - Samsun Kadın Doğum ve Çocuk Hastanesi, Samsun
  - Ondokuz Mayıs Üniversitesi Tıp Fakültesi, Samsun

IPD SHARING:
Plan to Share IPD: No